CLINICAL TRIAL: NCT06656871
Title: Biostimulants Application to Vegetables
Brief Title: Biostimulants Application to Lettuce
Acronym: SwE4WEEKS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Sara Baldassano, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SwE4WEEKS23
Record Dates: First submitted 2024-10-19; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2023-03

CONDITIONS: Nutrition, Healthy; Glucose Metabolism Disorders; Lipid Metabolism Disorders; Dietary Deficiency
MeSH Terms: conditions — Glucose Metabolism Disorders; Lipid Metabolism Disorders; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): The control group received lettuce (control lettuce 100 grams/day) that was without any biostimulation with Ecklonia Maxima algae but with the same characteristic of SwE lettuce (soil, water, harvesting time) for 4 weeks.
- Biostimulated SwE lettuce intervention group (Experimental): The SwE lettuce intervention group received lettuce biostimulated with Ecklonia Maxima algae (SwE lettuce, 100 grams/day) for 4 weeks
  Interventions: Dietary Supplement: Biostimulated lettuce supplementation
- Iron tablet intervention group (Experimental): The iron tablet intervention group received iron supplementation (30 mg, 1 tablet/day of iron) for 4 weeks
  Interventions: Dietary Supplement: iron supplementation

INTERVENTIONS:
Dietary Supplement: iron supplementation — The iron tablet group received iron supplementation (30 mg, 1 tablet/day of iron) for 4 weeks
  Arms: Iron tablet intervention group
Dietary Supplement: Biostimulated lettuce supplementation — the intervention group SwE lettuce group received lettuce biostimulated with Ecklonia Maxima algae (SwE lettuce, 100 grams/day) daily for 4 weeks
  Arms: Biostimulated SwE lettuce intervention group

SUMMARY:
Biostimulants application to vegetables is a useful agronomic approach to reduce the use of pesticides and to improve crop yield and quality by a naturally functionalizing process. The aim of the study is to verify the effects of a nutritional intervention with lettuce Biostimulated by application of seaweed extracts derived from Ecklonia maxima (SwE) in a healthy population in order to assess influence on specific essential minerals like calcium, potassium iron, magnesium, phosphorous (Primary outcome) and metabolisms like glucose, lipid, iron homeostasis (Secondary outcome).

DETAILED DESCRIPTION:
The present project aims to investigate the benefits of biostimulants lettuce in a cohort of healthy individuals. Biostimulants are organic and inorganic compounds or microorganisms that when applied to plants can enhance plants' growth, yield, and tolerance to stress. Seaweed extract treatment seems to enhance mineral concentration in crops. Participants will be fed with biostimulated lettuce or a tablet of iron daily in order to study the influence on hematological parameters.

A cohort of healthy subjects will be divided into a control group, receiving control lettuce, lettuce SwE group, receiving biostimulated lettuce and iron tablet group receiving iron bisglycinate (30 mg) supplement in tablet for a total of 4 weeks. Blood samples will be collected in specific tubes before (baseline) and after the nutritional intervention (T2). The group will eat 100 grams of Lettuce (control group) and 100 grams of SwE Biostimulated lettuce (intervention group lettuce) for 4 weeks (100 grams/daily) or a tablet of iron (intervention group iron tablet) and collect blood samples (serum and plasma) baseline, before starting the nutritional intervention and after 4 weeks (T2).

Each subject will be subjected to two venous blood samples taken at the beginning of the observation and at the end. The samples obtained will be transported in certified containers for the safe transport of biological samples, and, subsequently, processed by the experimenters at the laboratories of the Molecular Biology section of the University of Palermo. Serum and plasma will be obtained from each blood sample. All information thus obtained will be recorded in a database in which each person will be identified with a numerical code, in order to comply with current privacy regulations. Body weight, Barefoot standing height, Body mass index, Body composition will be measured in the different groups of study. Samples will be analyzed and compared for glucose, insulin, total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides, Ferritin, Iron, transferrin, Magnesium, Calcium, Potassium, Phosphate, Potassium.

Statistical analysis plan:

Student t tests will be used to compare the baseline characteristics of the groups. Changes between baseline and follow-up will be analyzed by one-way ANOVA followed by Sidak post test. A P < 0.05 will be considered to be statistically significant by using appropriate software.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 70 years
* Italian Ethnicity
* Body mass index between 18.5 and 28.5 kg/m2
* Clinically Healthy

Exclusion Criteria:

* Chronic disease
* Use of drugs
* Pregnancy
* Exogenous hormones
* Breastfeeding
* Use of supplements
* sensitivity to lettuce

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Measurement of minerals concentration in participants | 4 weeks
  Calcium (mg/dL), Phosphate (mg/dL), Magnesium (mg/dL) will be assessed in serum at baseline and after 4 weeks.
Measurement of iron concentration in participants | 4 weeks
  Iron (μg/dL) will be assessed in serum at baseline and after 4 weeks.
Measurement of Potassium concentration in participants | 4 weeks
  Potassium (mmol/L) will be assessed in serum at baseline and after 4 weeks.

SECONDARY OUTCOMES:
Measurement of ferritin in participants | 4 weeks
  Ferritin (ng/dL) will be measured in serum at baseline and after 4 weeks
Measurement of lipid metabolism markers in participants | 4 weeks
  triglicerises, HDL, LDL, cholesterol (in mg/dL) will be measured in serum at baseline and after 4 weeks
Measurement of insulin in participants | 4 weeks
  insulin (mUI/L) will be measured in serum at baseline and after 4 weeks
Measurement of transferrin in participants | 4 weeks
  transferrin (mg/dL) will be measured in serum at baseline and after 4 weeks
Measurement of % saturation of transferrin in participants | 4 weeks
  % saturation of transferrin will be measured in serum at baseline and after 4 weeks
Measurement of glucose in participants | 4 weeks
  glucose (mg/dL) will be measured in serum at baseline and after 4 weeks

OTHER OUTCOMES:
Measurement of Height in participants | 4 weeks
  Height (meters) will be assessed at baseline and after 4 weeks
Measurement of body mass index (BMI) in participants | 4 weeks
  weight in kilograms, height in meters will be aggregated to arrive at one reported value (weight and height will becombined to report BMI in kg/m^2).
Measurement of body weight in participants | 4 weeks
  Body weight (kg) will be assessed at baseline and after 4 weeks
Measurement of body composition in participants | 4 weeks
  lean mass as percent of body weight and fat mass as percent of body weight will be assessed at baseline and after 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- NABbio, STEBICEF department, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No
Because is forbidden by the Italian Low

REFERENCES:
- [Background] ttps://www.mdpi.com/2073-4395/12/6/1361 Description: Plant-Derived Biostimulants Differentially Modulate Primary and Secondary Metabolites and Improvethe Yield Potential of Red and Green Lettuce Cultivars
- [Derived] Di Gaudio F, Vasto S, Sabatino L, Ferrantelli V, Macaluso A, Caldarella R, Di Rosa L, Caldara GF, Proia P, Baldassano S. Consumption of lettuce with seaweed extract biostimulant application improved iron homeostasis in a randomized interventional trial of healthy individuals. Sci Rep. 2025 Mar 6;15(1):7799. doi: 10.1038/s41598-025-91380-7. PMID 40050333